CLINICAL TRIAL: NCT06953089
Title: A Phase II, Multicenter, Open-Label Trial of DB-1311 in Combination With BNT327 or DB-1305 in Participants With Advanced/Metastatic Solid Tumors
Brief Title: DB-1311 in Combination With BNT327 or DB-1305 in Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-1311-201
Record Dates: First submitted 2025-04-09; First posted 2025-05-01 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
Keywords: B7-H3; PD-L1/VEGF-A; TROP2 (Trophoblast cell surface antigen 2); ADC (antibody-drug conjugate); HNSCC (head and neck squamous cell carcinoma); HCC (hepatocellular carcinoma); Melanoma; NSCLC(non-small cell lung cancer); OC (ovarian cancer)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular; Melanoma; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 Cohort 1A, DB-1311/BNT324+ BNT327 combination therapy (Experimental): Escalating combination dose levels of DB-1311/BNT324 and BNT327 to define RP2D (Recommended Phase 2 Dose) and RP2D-1 in target population.
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327
- Part 1 Cohort 2, DB-1311/BNT324+ DB-1305 /BNT325 combination therapy (Experimental): Escalating combination dose levels of DB-1311/BNT324 and DB-1305/BNT325 to define RP2D and RP2D-1 in target population.
  Interventions: Drug: DB-1311/BNT324; Drug: DB-1305/BNT325
- Part 2 Arm 1: RP2D of DB-1311/BNT324 + BNT327 (Experimental): In participants with unresectable advanced/metastatic HCC
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327
- Part 2 Arm 2: RP2D of DB-1311/BNT324 + BNT327 (Experimental): In participants with unresectable advanced/ metastatic CC
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327
- Part2 Arm 3:RP2D of DB-1311/BNT324 + BNT327 (Experimental): In participants with unresectable advanced/metastatic melanoma
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327
- Part 2 Arm 4: RP2D of DB-1311/BNT324 + BNT327 and RP2D-1 of DB-1311/BNT324 + BNT327 (Experimental): In participants with recurrent/metastatic HNSCC
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327
- Part 2 Arm 5: RP2D of DB-1311/BNT324 +DB-1305/BNT325 and RP2D-1 of DB-1311/BNT324 +DB-1305/BNT325 (Experimental): In participants with advanced/unresectable metastatic NSCLC
  Interventions: Drug: DB-1311/BNT324; Drug: DB-1305/BNT325
- Part 1 Cohort 1B, DB-1311/BNT324+ BNT327 combination therapy (Experimental): Escalating combination dose levels of DB-1311/BNT324 and BNT327 to define RP2D and RP2D-1 in target population.
  Interventions: Drug: DB-1311/BNT324; Drug: BNT327

INTERVENTIONS:
Drug: DB-1311/BNT324 — Administered I.V.
Drug: BNT327 — Administered I.V.
  Arms: Part 1 Cohort 1A, DB-1311/BNT324+ BNT327 combination therapy; Part 1 Cohort 1B, DB-1311/BNT324+ BNT327 combination therapy; Part 2 Arm 1: RP2D of DB-1311/BNT324 + BNT327; Part 2 Arm 2: RP2D of DB-1311/BNT324 + BNT327; Part 2 Arm 4: RP2D of DB-1311/BNT324 + BNT327 and RP2D-1 of DB-1311/BNT324 + BNT327; Part2 Arm 3:RP2D of DB-1311/BNT324 + BNT327
Drug: DB-1305/BNT325 — Administered I.V.
  Arms: Part 1 Cohort 2, DB-1311/BNT324+ DB-1305 /BNT325 combination therapy; Part 2 Arm 5: RP2D of DB-1311/BNT324 +DB-1305/BNT325 and RP2D-1 of DB-1311/BNT324 +DB-1305/BNT325

SUMMARY:
A Phase II, Multicenter, Open-Label Trial of DB-1311 in combination with BNT327 or DB-1305 in Participants with Advanced/Metastatic Solid Tumors

DETAILED DESCRIPTION:
This is a phase II, multicenter, open-label, two-part trial designed to evaluate the safety and preliminary efficacy of DB-1311 in combination with BNT327 or DB-1311 in combination with DB-1305 in targeted participants.

Participants with recurrent, progressive as well as advanced, metastatic hepatocellular carcinoma (HCC), cervical cancer (CC), melanoma, head and neck squamous cell carcinoma (HNSCC), platinum-resistant ovarian cancer (PROC) or non-small cell lung cancer (NSCLC) are eligible to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years or acceptable age according to local regulations at the time of voluntarily signing informed consent.
* At least one measurable lesion as assessed by the Investigator according to RECIST v1.1 criteria.
* Has a life expectancy of ≥ 3 months.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
* Has adequate organ function within 7 days prior to enrollment/randomization,
* Has adequate treatment washout period prior to the first dose of trial treatment.

  * For HCC patients: Histological/cytological confirmed diagnosis of HCC or clinically confirmed diagnosis of HCC; Has a Child-Pugh class A liver score.
  * For CC patients: Has persistent, recurrent or metastatic cervical cancer with squamous cell, adenocarcinoma, or adenosquamous histology
  * For Melanoma patients: Histologically or cytologically confirmed diagnosis of unresectable Stage III or metastatic melanoma.
  * For PROC patients (Cohort A): Participants must have a confirmed diagnosis of OC, primary peritoneal cancer, or fallopian tube cancer, all of which with high-grade serous histology. Patients must have platinum-resistant disease.
  * For HNSCC patients: Histologically or cytologically confirmed recurrent (recurrent disease that is not amendable to curative treatment with local/ or systemic therapies)/ (disseminated) HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies.
  * For NSCLC patients: Pathologically documented Stage IIIB or IIIC NSCLC not amenable for radical surgery or definitive chemoradiation or Stage IV NSQ NSCLC. Not harboring an EGFR-sensitizing mutation or ALK gene rearrangements or other onco-driver gene mutations

Exclusion Criteria:

* 1. Prior treatment with B7H3 targeted therapy.
* Prior treatment with antibody-drug conjugate with topoisomerase inhibitor.
* Is a candidate to locoregional treatment with potential to induce complete or near complete response and prolonged tumor control, per investigator's assessment.
* Has an uncontrolled concomitant or intercurrent illness, that in the opinion of the investigator, contra-indicates trial participation, limits compliance with trial procedures or substantially increases the risk of incurring AEs.
* Has uncontrolled or significant cardiovascular disease. Has clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring drainage, peritoneal shunt, or cell-free concentrated ascites reinfusion therapy.
* Has a history of (non-infectious) ILD/pneumonitis.
* Any autoimmune, connective tissue or inflammatory disorders.
* Has spinal cord compression or clinically active central nervous system (CNS) metastases.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤1 or baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of participants with Dose Limiting Toxicities (DLTs). | During the DLT evaluation period, i.e., the time of initiation of the first dose of investigational medicinal product (IMP) up to 21 days
Part 1: Treatment-emergent adverse events (TEAEs) and treatment-emergent serious AE (TESAEs) | up to follow up period, e.g. up to 72 months.
Part 2: Treatment-emergent adverse events (TEAEs) and treatment-emergent serious AE (TESAEs) [By arm and dose level] | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 2: Objective response rate (ORR), defined as the proportion of participants in whom a confirmed Complete response (CR) or PR is observed as best overall response (per RECIST 1.1 based on the investigator's assessment)by arm and dose level. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months

SECONDARY OUTCOMES:
Part 1: ORR, defined as the proportion of participants in whom a confirmed CR or PR is observed as best overall response (per RECIST 1.1 based on the investigator's assessment). | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Duration of response (DoR) per RECIST 1.1 based on the investigator's assessment. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Overall survival (OS) | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Disease-control rate (DCR) per RECIST 1.1 based on the investigator's assessment. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Time to response (TTR) per RECIST 1.1 based on the investigator's assessment. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Progression-free survival (PFS) per RECIST 1.1 based on the investigator's assessment. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1: Cancer antigen 125 (CA-125) response rate assessed per Gynecological Cancer Intergroup (GCIG) criteria in participants with platinum-resistant ovarian cancer (PROC). | From the time of initiation of the first dose of IMP to end of Part 1
Part 1: Cancer antigen 125 (CA-125) response rate assessed per Gynecological Cancer Intergroup (GCIG) criteria in participants with PROC. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 2:Treatment-emergent adverse events (TEAEs) and treatment-emergent serious AE (TESAEs) | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Maximum observed concentration (Cmax) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with BNT327. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Maximum observed concentration (Cmax) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with DB-1305/BNT325. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Time to reach maximum observed concentration (Tmax) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with BNT327. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Time to reach maximum observed concentration (Tmax) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with DB-1305/BNT325. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with BNT327. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Area under the concentration-time curve from time 0 extrapolated to infinity (AUCinf) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with DB-1305/BNT325. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Terminal elimination half-life (t1/2) of DB-1311/BNT324 total ADC, total antibody and unconjugated P1021 in combination with BNT327. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Terminal elimination half-life (t1/2) of DB-1311/BNT324 ADC, total antibody and unconjugated P1021 in combination with DB-1305/BNT325. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and 2: Anti-drug antibody (ADA) prevalence: the proportion of participants who are ADA positive at any point in time (at baseline and post-baseline). | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months
Part 1 and Part 2: ADA incidence: the proportion of participants having treatment-emergent ADA. | From the time of initiation of the first dose of IMP to end of study, i.e., up to 72 months

CONTACTS AND LOCATIONS:
Locations (37):
- United States (15):
  - USA06-0, Los Angeles, California
  - USA16-0, Los Angeles, California
  - USA01-0, Wheat Ridge, Colorado
  - USA08-0, Florida City, Florida
  - USA10-0, Atlanta, Georgia
  - USA11-0, Bethesda, Maryland
  - USA14-0, Lincoln, Nebraska
  - USA04-0, New York, New York
  - USA15-0, Portland, Oregon
  - USA03-0, Charleston, South Carolina
  - USA13-0, Anderson, Texas
  - USA12-0, Houston, Texas
  - USA05-0, Virginia Beach, Virginia
  - USA09-0, Puyallup, Washington
  - USA07-0, Spokane, Washington
- Australia (4):
  - AUS07-0, North Sydney, New South Wales
  - AUS06-0, Benowa, Queensland
  - AUS04-0, Birtinya, Queensland
  - AUS05-0, Adelaide, South Australia
- China (16):
  - CHN02-0, Beijing, Beijing Municipality
  - CHN13-0, Beijing, Beijing Municipality
  - CHN23-0, Beijing, Beijing Municipality
  - CHN17-0, Dongguan, Guangdong
  - CHN06-0, Henan, Henan
  - CHN12-0, Xinxiang, Henan
  - CHN04-0, Hubei, Hubei
  - CHN26-0, Wuhan, Hubei
  - CHN34-0, Wuhan, Hubei
  - CHN11-0, Changsha, Hunan
  - CHN16-0, Xuzhou, Jiangsu
  - CHN35-0, Shenyang, Liaoning
  - CHN25-0, Xi'an, Shaanxi
  - CHN04-0, Shanghai, Shanghai Municipality
  - CHN01-0, Shanghai, Shanghai Municipality
  - CHN24-0, Chengdu, Sichuan
- Taiwan (2):
  - TWN01-0, Taipei, Taipei
  - TWN02-0, Taipei, Taipei

IPD SHARING:
Plan to Share IPD: Undecided